CLINICAL TRIAL: NCT02903745
Title: Knowledge Attitudes Beliefs and Practices Regarding HIV Among Teenagers in French Guiana
Acronym: CAPADO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: capado
Record Dates: First submitted 2016-09-06; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: HIV
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: observational

SUMMARY:
French Guiana is the French territory where the prevalence of HIV is highest. in order to determine the knowledge attitudes, beliefs, and practices among the target group of teenagers attending the public school system a survey was conducted in 2011. schools and classrooms were randomly selected, and a structured questionnaire was administered. Descriptive statistics were obtained and multivariate logistic regression was used to determine predictors of main outcomes such as age at first sex.

the results will be used to guide prevention of HIV and sexually transmitted infections though the school system.

ELIGIBILITY:
Inclusion Criteria:

* attending the public school system of french guiana

Exclusion Criteria:

* refusal to participate

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: randomly selected teenagers attending the public school system of french guiana
Sampling Method: Probability Sample
Enrollment: 1603 (Actual)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
knowledge, attitudes, behaviours, and practices relative to HIV/AIDS and sexually transmitted infections | when the interview was conducted
  a structured questionnaire was used. it was administered face to face with usually 5 possible responses. Scores were established using similar questions exploring related areas of HIV.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Cayenne, Cayenne, French Guiana, France